CLINICAL TRIAL: NCT03287986
Title: Brain Markers of Suicide Risk and Psychological Pain in Elderly Depressed Patients
Acronym: SPAD-IRM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2016/FJMW-01
Record Dates: First submitted 2017-04-21; First posted 2017-09-19 (Actual); Last update posted 2020-03-09 (Actual); Status verified 2020-03

CONDITIONS: Depressive Disorder; Suicide, Attempted
Keywords: Elderly; MRI
MeSH Terms: conditions — Depressive Disorder; Suicide, Attempted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — DNA, blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Suicide attempters: Depressed patients over 60 years of age with a personal history of suicide attempts scanned with MRI
  Interventions: Other: MRI
- Patient controls: depressed patients over 60 years of age without a personal history of suicide attempt scanned with MRI
  Interventions: Other: MRI
- Healthy Controls: Healthy subjects over 60 years, not depressed and without personal history of severe mental illness or suicide attempts, scanned with MRI
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — Structural and functional sequences

SUMMARY:
The main objective of this study is to show MRI functional and structural differences between depressed elderly patients with a history of attempted suicide compared to depressed elderly patients with no history of attempted suicide and to elderly subjects with no personal history of depression or attempted suicide (healthy controls).

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* be a member or beneficiary of a health insurance plan
* aged 60 years-old or more
* must be right-handed
* with a diagnosis of a current major depressive episode of moderate to severe severity according to diagnostic criteria.
* with or without a personal history of attempted suicide during life
* hospitalized or followed by a consultant in the department of Psychiatry of Nîmes University Hospital or in the Sophoras private clinic

Exclusion Criteria:

* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* under safeguard of justice
* refuses to sign the consent
* It is impossible to give the subject informed information
* Current psychotic symptoms.
* Bipolar disorder.
* The subject presents an acute somatic decompensation incompatible with the realization of this study.
* The patient presents a mental confusion or a known Mini Mental State Examination score <24.
* Central neurological disease known in particular degenerative pathology, severe cranial trauma and severe cerebrovascular disease.
* Schizophrenia and other known psychotic disorders.
* Electroconvulsive therapy in the 12 months prior to study
* Inability to perform neuropsychological tests because of a language problem, poor understanding, a major tremor, inability to sit still, a major sight problem that cannot be corrected, or other severe cognitive impairment
* Contra-indication to magnetic resonance imaging (MRI): ferromagnetic implant in the body, piercing, claustrophobia, inability to remain elongated for 45 minutes.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elderly depressed patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Brain functional activity during unfairness | Day 0
  Contrast in BOLD signal measured by 3T-Magnetic Resonance Imaging (MRI) during the fair vs unfair trials of the Ultimatum Game

SECONDARY OUTCOMES:
Brain structural volumes | Day 0
  T1 sequence measured by MRI in each participant
Brain structural connectivity | Day 0
  Diffusion Tensor Imaging measured by MRI in each participant
Brain functional connectivity | Day 0
  Resting state activity measured by MRI in each participant
Correlation of MRI measures with psychological pain measures | Day 0
  Psychological pain will be measured by the Visual Analog Scale (Olié et al. 2010) in each participant

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice Jollant, MD PhD, Principal Investigator — CHU Nîmes
Locations (1):
- CHU Nimes, Nîmes, France

IPD SHARING:
Plan to Share IPD: No